CLINICAL TRIAL: NCT02870478
Title: A Study of Time and Dose-dependent Effect of Low Concentration Atropine on Accommodation and Pupil Size
Brief Title: The Effects of Low Concentration Atropine on Pupil Size and Accommodation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IND 128961
Record Dates: First submitted 2016-07-27; First posted 2016-08-17 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.01% atropine daily (Active Comparator): Nightly dosing of 0.01% atropine
  Interventions: Drug: Atropine
- 0.01% atropine twice per week (Experimental): Atropine dosed twice per week
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Atropine — Dosing frequency comparison, using atropine sulfate 1% solution diluted to 0.01% and 0.05% by Leiter's Compounding Pharmacy
  Other Names: atropine sulfate ophthalmic solution

SUMMARY:
The purpose of this study is to determine whether less frequent dosing of atropine drops may be as effective as daily dosing for the treatment of progressive myopia.

DETAILED DESCRIPTION:
Myopia has become an epidemic in developed countries, particularly in Asian countries and in the United States. Myopia, or near-sightedness, is a result of uncontrolled axial elongation of the eye. Besides needing optical correction in order to see clearly, myopia can result in many sight-threatening complications, such as retinal thinning, retinal holes and tears, retinal detachment, and vascular proliferation. Atropine drops have been used in clinical practice for over 100 years at varying concentrations and different dosing regimens. The proposed small study seeks to establish evidence-based treatment (dosing) guidelines for the use of low dose atropine for myopia control.

The specific objectives of this study are:

1. To assess the effects of 0.01% atropine on pupil dilation and accommodation as a measure of active drug levels in the eye when dosed twice per week compared to daily
2. To assess the subjective effects of 0.01% atropine on the subjects' vision

The study will involve one 60-minute screening session, twenty 15-minute testing sessions, and one 8-hour testing session, for a total of 14 hours over five to six weeks. Following the screening exam (information will be collected on the screening form), the subject will be randomly assigned to treat their non-dominant eye with:

1. 0.01% daily dosing for two weeks followed by a 1-week washout then 0.01% twice per week for two weeks
2. 0.01% twice per week dosing for two weeks, followed by a 1-week washout, then 0.01% daily for two weeks.

Test sessions (expected to be no more than 15 mins in length) will be held daily during the testing period and scheduled at the subject's convenience. Session measurements will include best-corrected visual acuity, subjective amplitude of accommodation, objective amplitude of accommodation, and pupil size, as described previously (see screening section 7b). An anterior segment slit lamp biomicroscopy exam will also be performed to ensure good ocular health. The subject will also be asked to fill out a brief symptom questionnaire (attached) while they are present for the test session. Information will be recorded on the data collection sheet for this portion of the testing.

Additionally, measurements of pupil size and accommodation will be taken prior to the instillation of a single dose of 0.01% atropine, and then at 1min, 5 min, 30 min, 1hr, 2hr, 4hr, and 8hr post-instillation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have vision that is correctable to 20/20 in each eye
* Participants must also have normal binocular vision (no history of manifest eye turns or eye surgeries to correct an eye turn)
* Participants must have normal accommodation (amplitude and facility within a normal range based on the subject's age)
* Participants must have normal ocular health

Exclusion Criteria:

* Previous chronic use of atropine
* Participants who are pregnant, plan to become pregnant, or are breastfeeding
* Sensitivity or allergy to atropine

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-07; Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Change in pupil size at 1 week | Measured at baseline and again 1 week after first using drop

CONTACTS AND LOCATIONS:
Overall Officials: Maria Liu, OD, MPH, PhD, Principal Investigator — UC Berkeley
Locations (1):
- UC Berkeley, Department of Vision Science, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Undecided